CLINICAL TRIAL: NCT03500627
Title: A Phase 1 Open-Label Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of OP-101 (Dendrimer N-Acetyl-Cysteine) After Intravenous Administration in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of OP-101 After Intravenous Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orpheris, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OP-101-002
Record Dates: First submitted 2018-03-27; First posted 2018-04-18 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Adrenoleukodystrophy (ALD); Childhood Cerebral Adrenoleukodystrophy (ccALD); OP-101; Dendrimer; N-Acetyl-Cysteine (NAC)
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 20 mg/kg OP-101 administered intravenously for over 1 hour.
  Interventions: Drug: OP-101
- Cohort 2 (Experimental): 40 mg/kg OP-101 administered intravenously for over 1 hour.
  Interventions: Drug: OP-101
- Cohort 3 (optional) (Experimental): 80 mg/kg OP-101 administered intravenously for over 1 hour.
  Interventions: Drug: OP-101

INTERVENTIONS:
Drug: OP-101 — Intravenous Injection of OP-101 in healthy volunteers.

SUMMARY:
A clinical study to measure the effect of OP-101 after being administered intravenously in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 32 kg/m^2.
* Is in general good health, based upon the results of a medical history assessment, physical examination, vital signs, laboratory profile, and 12-lead electrocardiogram (ECG), as judged by the investigator.
* Female subjects may not be pregnant, lactating, or breastfeeding.
* Subjects must have a negative urine test for drugs of abuse, cotinine, and breath alcohol test at screening and Check-in.

Key Exclusion Criteria:

* Evidence of clinically significant hematologic, renal, endocrine, pulmonary, cardiac, gastrointestinal, hepatic, psychiatric, neurologic, immunologic, allergic disease, or any other condition that, in the opinion of the Investigator, might significantly interfere with the absorption, distribution, metabolism, or excretion of study drug, or place the subject at an unacceptable risk as a participant in this study.
* History of malignancy (other than successfully treated basal cell or squamous cell skin cancer).
* History or presence of an abnormal ECG that, in the opinion of the Investigator, is clinically significant.
* Has used any product containing nicotine within 90 days prior to screening or intends to use any product containing nicotine during the course of the study.
* Has used medications that affect gastrointestinal motility or gastric emptying; such as metoclopramide, proton pump inhibitors, and H2 blockers; within 30 days prior to Day 1.
* Has used prescription or over-the-counter medication, vitamins/herbal supplements (with the exception of hormonal contraceptives) within 14 days prior to Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events Graded as Assessed by CTCAE Version 4.0 | Screening to Day 15.
  Evaluate the safety and tolerability of OP-101 after single IV doses in healthy subjects by monitoring and documenting all adverse events, which include laboratory test variables.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Profile Analysis | Days 1, 2, 3, 4, 8, and 15.
  Determine the PK profile of OP-101 after single IV doses in healthy subjects as determined by plasma concentrations using the PK Concentration Population.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, MD, Study Chair — Orpheris, Inc.
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States